CLINICAL TRIAL: NCT05251701
Title: Personal KinetiGraph® Clinical Validation Study
Status: Completed | Type: Observational
Sponsor: Global Kinetics Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: Study 006
Record Dates: First submitted 2021-10-29; First posted 2022-02-23 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-09

CONDITIONS: Movement Disorders; Parkinson Disease
MeSH Terms: conditions — Movement Disorders; Parkinson Disease | interventions — Drug Delivery Systems

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: Personal KinetiGraph® (PKG®) System — The PKG® System includes a wrist-worn device that records and measures movement patterns in conditions such as Parkinson's disease.

SUMMARY:
The purpose of this study is to clinically validate new measures of the Personal KinetiGraph® (PKG®).

DETAILED DESCRIPTION:
This is a prospective, observational research study of the Personal KinetiGraph (PKG) System. The PKG System is intended to quantify kinematics of movement disorder symptoms in conditions such as Parkinson's disease, including tremor, bradykinesia and dyskinesia. This study aims to clinically validate new PKG assessments such as walking, Device Assisted Therapy readiness, Percent Time Bradykinesia, Percent Time Dyskinesia, fall prediction, disease progression and non-motor. The clinical validation will require enrollment of both subjects with a diagnosis of movement disorder, such as Parkinson's disease, and healthy control subjects who do not a neurological disorder.

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to sign a written informed consent for study participation
* Existing diagnosis of a movement disorder or a healthy control subject without diagnosis of a movement disorder

Exclusion Criteria:

* Bedridden, wheelchair confined, or requires the regular use of an assistive gait device (e.g., walker, cane, etc.)
* Occupation that involves repetitive movement or complete immobility (e.g., janitor, construction, or sedentary with no/limited arm movements such as a taxi driver)
* In the investigator's or sponsor's opinion, subject has any unstable or clinically significant condition that would impair the participant's ability to complete the required PKG watch wear (e.g., subject unable to complete PKG wear instructions per Patient Instruction Manual), complete required assessments or interfere with data collection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects will be identified from routine clinical care
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2022-12-09 (Actual); Primary Completion 2023-08-16 (Actual); Study Completion 2025-09-03 (Actual)

PRIMARY OUTCOMES:
Evaluation of new PKG assessments to be clinically validated for Gait/walking using movement data collected from the PKG Watch | 2-3 years
  The PKG's step detection system and manual step counts may be compared between healthy controls and person's with Parkinson's disease, while their walking is video recorded.
Evaluation of new PKG assessments to be clinically validated for Device Assisted Therapy readiness using movement data collected from the PKG Watch | 2-3 years
  For this outcome, patients may be classified as Device Assisted Therapy (DAT) criteria positive or criteria negative. DAT readiness may be evaluated using the Movement Disorder Society-Sponsored Unified Parkinson's Disease Rating Scale (MDS-UPDRS). The MDS-UPDRS evaluates motor and non-motor symptoms in persons with Parkinson's and consists of 4 parts. Parts I and II each contain 13 questions, Part III contains 33 and Part IV contains 6. Each score ranges from 0 (normal) to 4 (severe). Higher scores indicate a greater impact of Parkinson's disease symptoms. PKG measurements may be compared to the patient's clinical characteristics and MDS-UPDRS scores.
Evaluation of new PKG assessments to be clinically validated for Percent Time Bradykinesia using movement data collected from the PKG Watch (PTB) | 2-3 years
  Data collected from the PKG system may be compared to scores from the Movement Disorder Society-Sponsored Unified Parkinson's Disease Rating Scale (MDS-UPDRS) and the Parkinson's Disease Questionnaire (PDQ-39). The MDS-UPDRS evaluates motor and non-motor symptoms in persons with Parkinson's and consists of 4 parts. Parts I and II each contain 13 questions, Part III contains 33 and Part IV contains 6. Each score ranges from 0 (normal) to 4 (severe). Higher scores indicate a greater impact of Parkinson's disease symptoms. The PDQ-39 includes 39 questions that assess Parkinson's disease health related quality of life. Each dimension total score range from 0 (never have difficulty) to 100 (always have difficulty).
Evaluation of new PKG assessments to be clinically validated for Percent Time Dyskinesia (PTD) using movement data collected from the PKG Watch | 2-3 years
  Data collected from the PKG system may be compared to scores from the Movement Disorder Society-Sponsored Unified Parkinson's Disease Rating Scale (MDS-UPDRS) and the Parkinson's Disease Questionnaire (PDQ-39). The MDS-UPDRS evaluates motor and non-motor symptoms in persons with Parkinson's and consists of 4 parts. Parts I and II each contain 13 questions, Part III contains 33 and Part IV contains 6. Each score ranges from 0 (normal) to 4 (severe). Higher scores indicate a greater impact of Parkinson's disease symptoms. The PDQ-39 includes 39 questions that assess Parkinson's disease health related quality of life. Each dimension total score range from 0 (never have difficulty) to 100 (always have difficulty).
Evaluation of new PKG assessments to be clinically validated for fall prediction using movement data collected from the PKG Watch | 2-3 years
  PKG measurements may be compared to data collected from freezing of gait questionnaire (FOG-Q) and posture analysis. The FOG-Q assesses freezing of gait severity and consists of 4 questions, each scored from 0-4. Higher scores indicates more severe freezing of gait. Step count performance may also be used to evaluate fall prediction. The PKG's step detection system and manual step counts may be compared between healthy controls and person's with Parkinson's disease, while their walking is video recorded.
Evaluation of new PKG assessments to be clinically validated for disease progression using movement data collected from the PKG Watch | 2-3 years
  Disease progression may be evaluated by predicting the levodopa response using severity levels of the Bradykinesia Score (BKS) and early morning Bradykinesia. Changes in PKG measurements may be compared to the MDS-UPDRS which evaluates motor and non-motor symptoms in persons with Parkinson's and consists of 4 parts. Parts I and II each contain 13 questions, Part III contains 33 and Part IV contains 6. Each score ranges from 0 (normal) to 4 (severe). Higher scores indicate a greater impact of Parkinson's disease symptoms.
Evaluation of new PKG assessments to be clinically validated for non-motor outcomes using non-motor scales | 2-3 years
  PKG system data may be compared to non-motor assessments such as the non-motor questionnaire (NMSQ). The NMSQ includes questions regarding non-motor symptoms such as difficulty swallowing, constipation, difficulty sleeping, cognition, mood. Higher scores indicate more non-motor symptoms.

SECONDARY OUTCOMES:
Evaluation of PKG scores to assess differences by age category | 2-3 years
  PKG measurements will be recorded and compared across age ranges (40-90 years old as defined in the Inclusion Criteria) for subjects enrolled. Age categories from 40-59 years old, 60-79 years old and 80-90 years old will be evaluated.
To compare PKG scores to standard Parkinson's disease assessments such as the Movement Disorder Specialist Unified Parkinson's Disease Scale | 2-3 years
  The MDS-UPDRS evaluates motor and non-motor symptoms in persons with Parkinson's and consists of 4 parts. Parts I and II each contain 13 questions, Part III contains 33 and Part IV contains 6. Each score ranges from 0 (normal) to 4 (severe). Higher scores indicate a greater impact of Parkinson's disease symptoms.
To compare PKG scores to standard Parkinson's disease assessments such as Parkinson's Disease Questionnaire (PDQ-39) | 2-3 years
  The PDQ-39 includes 39 questions that assess Parkinson's disease health related quality of life. Each dimension total score range from 0 (never have difficulty) to 100 (always have difficulty).
To compare PKG scores to standard Parkinson's disease assessments such as the Freezing of Gait Questionnaire (FOG-Q) | 2-3 years
  The FOG-Q assesses freezing of gait severity and consists of 4 questions, each scored from 0-4. Higher scores indicates more severe freezing of gait.
To compare PKG scores to standard Parkinson's disease assessments such as The Essential Tremor Rating Assessment Scale (TETRAS) | 2-3 years
  TETRAS assesses essential tremor severity and its impact on activities of daily living (ADL). The ADL section includes 12 items and the performance section includes 9. Each item is rated 0-4. Higher scores indicate more severe impacts of ADL and tremor.
To compare PKG scores to subject diaries | 2-3 years
  Subject diaries will include recordings of medication times, falls, symptoms and sleep.
To compare PKG scores to non-motor assessments such as the Non-Motor Symptoms Questionnaire (NMSQ) | 2-3 years
  The NMSQ includes 30 questions, answered either yes or no, and assesses the presence, not severity, of non-motor symptoms.
To compare PKG scores to sleep assessments such as Epworth Sleepiness Scale (ESS) and Parkinson's Disease Sleep Scale (PDSS) | 2-3 years
  The ESS includes 8 questions each scored from 0-3 with a maximum score of 24. The higher the ESS score, the higher that person's average sleep propensity or 'daytime sleepiness'.
  The PDSS includes 15 questions, each rated from 0 to 10, with 0 being "Awful" or "Always" and 10 being "Excellent" or "Never".
To compare PKG scores to the Montreal Cognitive Assessment (MoCA) | 2-3 years
  The MoCA is an assessment used for detecting cognitive impairment. The scores range from 0 to 30 with 0 being the lowest and 30 being the highest.
To compare PKG scores to quality of life measurements such as EuroQual 5-D (EQ-5D) | 2-3 years
  The EQ-5D assesses health-related quality of life. Each question is scored from either 1-3 or 1-5, with 1 indicating no problems and 3 or 5 indicating extreme problems.
To evaluate product usability and satisfaction for PKG Watch, docking station and PKG Portal | 2-3 years
  PKG product usability and satisfaction questionnaires will be used to evaluate this outcome. Responses to questions range from very difficult to very easy, strongly disagree to strongly agree, very uncomfortable to very comfortable.

CONTACTS AND LOCATIONS:
Overall Officials: Zoltan Mari, MD, Principal Investigator — Z Neurosciences, LLC.
Locations (1):
- Tucson Neuroscience Research, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: Undecided
Any clinical study IPD may be made available to other researchers including PKG data; demographics, such as age, gender, ethnicity; medical history, such as comorbid conditions and movement disorder history. Subject data will not include any personally identifiable information.

REFERENCES:
- [Background] Griffiths RI, Kotschet K, Arfon S, Xu ZM, Johnson W, Drago J, Evans A, Kempster P, Raghav S, Horne MK. Automated assessment of bradykinesia and dyskinesia in Parkinson's disease. J Parkinsons Dis. 2012;2(1):47-55. doi: 10.3233/JPD-2012-11071. PMID 23939408
- [Background] Horne MK, McGregor S, Bergquist F. An objective fluctuation score for Parkinson's disease. PLoS One. 2015 Apr 30;10(4):e0124522. doi: 10.1371/journal.pone.0124522. eCollection 2015. PMID 25928634
- [Background] Kotschet K, Johnson W, McGregor S, Kettlewell J, Kyoong A, O'Driscoll DM, Turton AR, Griffiths RI, Horne MK. Daytime sleep in Parkinson's disease measured by episodes of immobility. Parkinsonism Relat Disord. 2014 Jun;20(6):578-83. doi: 10.1016/j.parkreldis.2014.02.011. Epub 2014 Feb 24. PMID 24674770
- [Background] Braybrook M, O'Connor S, Churchward P, Perera T, Farzanehfar P, Horne M. An Ambulatory Tremor Score for Parkinson's Disease. J Parkinsons Dis. 2016 Oct 19;6(4):723-731. doi: 10.3233/JPD-160898. PMID 27589540

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-06-23): https://cdn.clinicaltrials.gov/large-docs/01/NCT05251701/Prot_SAP_000.pdf